CLINICAL TRIAL: NCT05425745
Title: A Placebo-Controlled, Double-Blind, Randomized, Phase 3 Study to Evaluate the Effect of 10 mg Obicetrapib in Participants With a History of HeFH Who Are Not Adequately Controlled by Their Lipid Modifying Therapies
Brief Title: Evaluate the Effect of Obicetrapib in Patients With HeFH on Top of Maximum Tolerated Lipid-Modifying Therapies.
Acronym: BROOKLYN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-8995-301
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Dyslipidemias; High Cholesterol; Hypercholesterolemia; Familial Hypercholesterolemia; Lipid Metabolism Disorder; Metabolic Disease; Lipid Metabolism, Inborn Errors; Genetic Disease, Inborn; Hyperlipoproteinemias
Keywords: Obicetrapib; BROOKLYN; Cholesteryl ester transfer protein (CETP) inhibitor; Heterozygous Familial Hypercholesterolemia (HeFH); LDL-C
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Hyperlipoproteinemia Type II; Lipid Metabolism Disorders; Metabolic Diseases; Lipid Metabolism, Inborn Errors; Genetic Diseases, Inborn; Hyperlipoproteinemias

STUDY DESIGN:
Intervention Model Description: Placebo-Controlled, double-blind, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo tablet made to resemble active
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): one placebo tablet once daily
  Interventions: Drug: Placebo
- Obicetrapib 10 mg (Experimental): one 10 mg Obicetrapib tablet once daily
  Interventions: Drug: Obicetrapib

INTERVENTIONS:
Drug: Obicetrapib — 10 mg Obicetrapib tablet
  Other Names: CETP-inhibitor
  Arms: Obicetrapib 10 mg
Drug: Placebo — placebo tablet made to resemble active
  Arms: Placebo

SUMMARY:
This study will be a placebo-controlled, double-blind, randomized, phase 3 study to Evaluate the Efficacy, Safety, and Tolerability of Obicetrapib in Participants with a History of Heterozygous Familial Hypercholesterolemia (HeFH).

DETAILED DESCRIPTION:
This study will be a placebo-controlled, double-blind, randomized, phase 3 study in participants with HeFH to evaluate the efficacy, safety, and tolerability of obicetrapib as an adjunct to diet and maximally tolerated lipid-lowering therapy. The screening period for this study will take up to 14 days. Afterwards, patients will be randomized to placebo or 10 mg obicetrapib for an 365-day treatment period. After the treatment period, participants will have an end-of-study follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of heterozygous familial hypercholesterolemia (HeFH) by 1) Genotyping (not a screening assessment), WHO Criteria/Dutch Lipid Clinical Network Criteria with a score of > 8 points; and/or Simon Broome Register Diagnostic Criteria for definite or possible Familial Hypercholesterolemia (FH)
* Maximally tolerated lipid Modifying therapy for at least 8 weeks prior to screening such as: ATV (40 or 80), or (ROS 20 or 40 mg), Ezetimide, Bempedoic Acid, PCSK9 targeted therapy for at least 4 doses
* Fasting serum LDL-C ≥70 mg/dL (≥1.80 mmol/L)

Exclusion Criteria:

* New York Heart Association class II or IV heart failure or last known left ventricular ejection fraction < 30%;
* Hospitalized for heart failure within 5 years prior to Screening
* Major adverse cardiac event (MACE) within 3 months prior to Screening;
* HbA1c ≥10%, or fasting glucose
* Formal diagnosis of homozygous familial hypercholesterolemia (HoFH)
* Uncontrolled severe hypertension, defined as either systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥100 mmHg prior to Randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ditmarsch, Study Director — NewAmsterdam Pharma
Locations (96):
- United States (20):
  - Site 01022, Jonesboro, Arkansas
  - Site 01015, Toluca Lake, California
  - Site 01009, Sarasota, Florida
  - Site 01023, Boise, Idaho
  - Site 01018, Chicago, Illinois
  - Site 01012, Iowa City, Iowa
  - Site 01007, Baton Rouge, Louisiana
  - Site 01005, Port Gibson, Mississippi
  - Site 01006, St Louis, Missouri
  - Site 01011, Lincoln, Nebraska
  - Site 01004, Norfolk, Nebraska
  - Site 01002, Morristown, New Jersey
  - Site 01010, New Providence, New Jersey
  - Site 01001, North Massapequa, New York
  - Site 01020, Morganton, North Carolina
  - Site 01019, Winston-Salem, North Carolina
  - Site 01008, Chattanooga, Tennessee
  - Site 01016, El Paso, Texas
  - Site 01013, Houston, Texas
  - Site 01014, Suffolk, Virginia
- Canada (9):
  - Site 06007, Brampton
  - Site 06008, Chicoutimi
  - Site 06005, Halifax
  - Site 06003, Montreal
  - Site 06009, Montreal
  - Site 06004, Québec
  - Site 06006, Sherbrooke
  - Site 06001, Vancouver
  - Site 06002, Victoria
- Czechia (6):
  - Site 02006, Brno
  - Site 02002, Hradec Králové
  - Site 02003, Prague
  - Site 02005, Prague
  - Site 02004, Prague
  - Site 02001, Uherské Hradiště
- Georgia (10):
  - Site 022001, Batumi
  - Site 022003, Tbilisi
  - Site 022004, Tbilisi
  - Site 022010, Tbilisi
  - Site 022006, Tbilisi
  - Site 022007, Tbilisi
  - Site 022008, Tbilisi
  - Site 022002, Tbilisi
  - Site 022005, Tbilisi
  - Site 022009, Tbilisi
- Netherlands (6):
  - Site 04001, Amsterdam
  - Site 04003, Arnhem
  - Site 04002, Deventer
  - Site 04004, Eindhoven
  - Site 04005, Roosendaal
  - Site 04006, Rotterdam
- Norway (2):
  - Site 023003, Bodø
  - Site 023002, Oslo
- Poland (5):
  - Site 05002, Bialystok
  - Site 05003, Lodz
  - Site 05004, Lodz
  - Site 05005, Zabrze
  - Site 05001, Zamość
- South Africa (9):
  - Site 018001, Bloemfontein
  - Site 018002, Cape Town
  - Site 018009, Centurion
  - Site 018006, Centurion
  - Site 018004, Parow
  - Site 018003, Somerset West
  - Site 018005, Somerset West
  - Site 018007, Tongaat
  - Site 018008, Umhlanga
- Spain (18):
  - Site 17004, A Coruña
  - Site 017001, Barcelona
  - Site 17002, Barcelona
  - Site 17003, Córdoba
  - Site 17018, Figueras
  - Site 17011, Granada
  - Site 17017, Huelva
  - Site 17012, Huesca
  - Site 17008, Las Palmas de Gran Canaria
  - Site 17010, Madrid
  - Site 17016, Madrid
  - Site 17007, Málaga
  - Site 17013, Sabadell
  - Site 17015, Santiago de Compostela
  - Site 17009, Seville
  - Site 17006, Seville
  - Site 17014, Valencia
  - Site 17005, Zaragoza
- United Kingdom (11):
  - Site 014006, Birmingham
  - Site 014012, Bristol
  - Site 014009, Cardiff
  - Site 014010, Chichester
  - Site 014001, Dundee
  - Site 014002, London
  - Site 014003, Manchester
  - Site 014008, Metropolitan Borough of Wirral
  - Site 014011, Penzance
  - Site 014005, Stevenage
  - Site 014004, West Bromwich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicholls SJ, Nelson AJ, Ditmarsch M, Kastelein JJP, Ballantyne CM, Ray KK, Navar AM, Nissen SE, Goldberg AC, Brunham LR, Curcio D, Wuerdeman E, Neild A, Kling D, Hsieh A, Dicklin MR, Ference BA, Laufs U, Banach M, Mehran R, Catapano AL, Davidson MH. Obicetrapib on top of maximally tolerated lipid-modifying therapies in participants with or at high risk for atherosclerotic cardiovascular disease: rationale and designs of BROADWAY and BROOKLYN. Am Heart J. 2024 Aug;274:32-45. doi: 10.1016/j.ahj.2024.05.002. Epub 2024 May 4. PMID 38705341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 513 patients were screened: out of 513, 354 participants were randomized: 236 participants to the obicetrapib 10 mg group and 118 participants to the placebo group
Period: Overall Study
Arm/Group | Placebo | Obicetrapib 10 mg
Started | 118 | 236
Completed | 110 | 226
Not Completed | 8 | 10
Not completed — Withdrawal of Consent | 3 | 3
Not completed — Death | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Did not return for end of study visit | 0 | 1
Not completed — End of study visit completed by phone | 1 | 0
Not completed — Subject decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Population is defined as all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Obicetrapib 10 mg | Total
Number analyzed (Participants) | 118 | 236 | 354
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (11.06) | 57 (12.70) | 56.9 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 125 | 190
  Male | 53 | 111 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 8 | 10
  Not Hispanic or Latino | 114 | 226 | 340
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 110 | 219 | 329
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 4 | 5
Baseline Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] — Baseline LDL-C is defined as the last measurement prior to the first dose of study drug. LDL-C was measured by Preparative Ultracentrifugation (PUC). Population: 4 participants were missing baseline LDL-C (measured by PUC). 2 pts baseline LDL-C results were not available due to low volume or hemolysis. 2 pts were randomized but did not receive study drug. Therefore, baseline values (baseline defined as the last measurement prior to the first dose of study drug) were not available.
  mg/dL
    number analyzed (Participants) | 118 | 232 | 350
    (all) | 119.9 (54.47) | 123.4 (49.23) | 121.65 (51.85)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 84 [PUC]
Description: LS mean percent change from baseline to Day 84 in Low-Density Lipoprotein Cholesterol (LDL-C) in the obicetrapib group compared to the placebo group [PUC]. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 84 Days
Population: Baseline Population is defined as all participants who were randomized in the study. Baseline values were defined as last measurement prior to the first dose of study drug. 2 participants in the obi arm were randomized but did not receive study drug, therefore the "n" for the obi arm baseline values did not exceed n=234. In addition, participants needed available labs at both baseline and Day 84.
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 232
percent change from baseline | .25 (2.480) | -36.05 (1.769)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -36.31, 95% CI 2-sided [-42.22 to -30.39], Standard Error of Mean 3.019

2. Secondary Outcome: Percent Change in Low Density Lipoprotein-Cholesterol (LDL-C) From Baseline to Day 180 [Martin/Hopkins]
Description: LS mean percent change from baseline to Day 180 in Low-Density Lipoprotein Cholesterol (LDL-C) in the obicetrapib group compared to the placebo group [Martin/Hopkins]. LDL-C value was calculated using the Martin/Hopkins equation unless TG >= 400 mg/dL or LDL-C <= 50 mg/dL; where, LDL-C value was measured directly by preparative ultracentrifugation (PUC).
Time Frame: 180 Days
Population: Baseline Population is defined as all participants who were randomized in the study. Baseline values were defined as last measurement prior to the first dose of study drug. 2 participants in the obi arm were randomized but did not receive study drug, therefore the "n" for the obi arm baseline values did not exceed n=234. In addition, participants needed available labs at both baseline and Day 180.
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 5.98 (2.925) | -31.80 (2.054)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -37.78, 95% CI 2-sided [-44.79 to -30.78], Standard Error of Mean 3.572

3. Secondary Outcome: Percent Change in Low Density Lipoprotein-Cholesterol (LDL-C) From Baseline to Day 365 [PUC]
Description: LS mean percent change from baseline to Day 365 in Low-Density Lipoprotein Cholesterol (LDL-C) in the obicetrapib group compared to the placebo group [PUC]. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 365 Days
Population: Baseline Population is defined as all participants who were randomized in the study. Baseline values were defined as last measurement prior to the first dose of study drug. 2 participants in the obi arm were randomized but did not receive study drug, therefore the "n" for the obi arm baseline values did not exceed n=234. In addition, participants needed available labs at both baseline and Day 365.
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 232
percent change from baseline | 10.30 (4.222) | -31.14 (2.544)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA — The hierarchical testing procedure would only be conducted if the previous secondary efficacy endpoint reached a statistically significant treatment effect at p-value<0.05; Least Squares (LS) Means = -41.45, 95% CI 2-sided [-51.14 to -31.76], Standard Error of Mean 4.938

4. Secondary Outcome: Percent Change in Apolipoprotein B (ApoB) From Baseline to Day 84
Description: LS mean percent change from baseline to Day 84 in apolipoprotein B (ApoB) in obicetrapib group compared to the placebo group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 2.93 (1.758) | -21.45 (1.219)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = -24.39, 95% CI 2-sided [-28.58 to -20.20], Standard Error of Mean 2.136

5. Secondary Outcome: Percent Change in Apolipoprotein B (ApoB) From Baseline to Day 180
Description: LS mean percent change from baseline to Day 180 in apolipoprotein B (ApoB) in obicetrapib group compared to the placebo group
Time Frame: 180 Days
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 6.02 (2.127) | -18.30 (1.472)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = -24.32, 95% CI 2-sided [-29.38 to -19.25], Standard Error of Mean 2.583

6. Secondary Outcome: Percent Change in Apolipoprotein B (ApoB) From Baseline to Day 365
Description: LS mean percent change from baseline to Day 365 in apolipoprotein B (ApoB) in obicetrapib group compared to the placebo group
Time Frame: 365 Days
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 8.15 (2.633) | -17.62 (1.663)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = -25.77, 95% CI 2-sided [-31.88 to -19.67], Standard Error of Mean 3.114

7. Secondary Outcome: Percent Change in Non-HDL-C From Baseline to Day 84
Description: LS mean percent change from baseline to Day 84 in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) in obicetrapib group compared to the placebo group
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 2.83 (2.188) | -31.62 (1.520)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = -34.45, 95% CI 2-sided [-39.67 to -29.24], Standard Error of Mean 2.661

8. Secondary Outcome: Percent Change in Non-HDL-C From Baseline to Day 180
Description: LS mean percent change from baseline to Day 180 in Non-high-density Lipoprotein Cholesterol (non-HDL-C) in obicetrapib group compared to the placebo group
Time Frame: 180 Days
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 5.92 (2.658) | -27.08 (1.855)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = -33.00, 95% CI 2-sided [-39.36 to -26.65], Standard Error of Mean 3.241

9. Secondary Outcome: Percent Change in Non-HDL-C From Baseline to Day 365
Description: LS mean percent change from baseline to Day 365 in Non-high-density Lipoprotein Cholesterol (non-HDL-C) in obicetrapib group compared to the placebo group
Time Frame: 365 Days
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 11.64 (3.905) | -25.84 (2.305)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA — The hierarchical testing procedure would only be conducted if the previous secondary efficacy endpoint reached a statistically significant treatment effect at p-value <0.05; Least Squares (LS) Means = -37.48, 95% CI 2-sided [-46.38 to -28.58], Standard Error of Mean 4.535

10. Secondary Outcome: Percent Change in HDL-C From Baseline to Day 84
Description: LS mean percent change from baseline to Day 84 in High-density Lipoprotein Cholesterol (HDL-C) in obicetrapib group compared to the placebo group
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 1.26 (5.078) | 139.92 (3.614)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 9, analysis 1]; Least Squares (LS) Means = 138.66, 95% CI 2-sided [126.42 to 150.90], Standard Error of Mean 6.244

11. Secondary Outcome: Percent Change in HDL-C From Baseline to Day 180
Description: LS mean percent change from baseline to Day 180 in High-density Lipoprotein Cholesterol (HDL-C) in obicetrapib group compared to the placebo group
Time Frame: 180 Days
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 2.63 (5.484) | 133.83 (3.730)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 9, analysis 1]; Least Squares (LS) Means = 131.20, 95% CI 2-sided [118.27 to 144.13], Standard Error of Mean 6.595

12. Secondary Outcome: Percent Change in HDL-C From Baseline to Day 365
Description: LS mean percent change from baseline to Day 365 in High-density Lipoprotein Cholesterol (HDL-C) in obicetrapib group compared to the placebo group
Time Frame: 365 Days
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 6.28 (5.994) | 127.67 (4.222)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 9, analysis 1]; Least Squares (LS) Means = 121.39, 95% CI 2-sided [107.02 to 135.76], Standard Error of Mean 7.333

13. Secondary Outcome: Percent Change in Lp(a) From Baseline to Day 84
Description: LS mean percent change from baseline to Day 84 in Lipoprotein (a) [Lp(a)] in obicetrapib group compared to the placebo group
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 10.52 (9.413) | -35.42 (4.527)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = -45.94, 95% CI 2-sided [-65.88 to -26.00], Standard Error of Mean 10.140

14. Secondary Outcome: Percent Change in Lp(a) From Baseline to Day 365
Description: LS mean percent change from baseline to Day 365 in Lipoprotein (a) [Lp(a)] in obicetrapib group compared to the placebo group
Time Frame: 365 Days
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 24.37 (37.111) | -29.93 (11.224)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p = 0.1648, ANCOVA — The hierarchical testing procedure would only be conducted if the previous secondary efficacy endpoint reached a statistically significant treatment effect at p-value<0.05; therefore hierarchical testing was stopped for subsequent secondary endpoints; Least Squares (LS) Means = -54.30, 95% CI 2-sided [-131.13 to 22.53], Standard Error of Mean 38.924

15. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Day 84
Description: LS mean percent change from baseline to Day 84 in Total Cholesterol (TC) in obicetrapib group compared to the placebo group
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 2.34 (1.796) | 12.09 (1.268)

16. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Day 180
Description: LS mean percent change from baseline to Day 180 in Total Cholesterol in obicetrapib group compared to the placebo group
Time Frame: 180 Days
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 4.44 (2.043) | 14.43 (1.438)

17. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Day 365
Description: LS mean percent change from baseline to Day 365 in Total Cholesterol in obicetrapib group compared to the placebo group
Time Frame: 365 Days
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 9.32 (2.801) | 13.92 (1.684)

18. Secondary Outcome: Percent Change in Triglycerides From Baseline to Day 84
Description: LS mean percent change from baseline to Day 84 in Triglycerides in obicetrapib group compared to the placebo group
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 10.16 (4.207) | -1.57 (2.580)

19. Secondary Outcome: Percent Change in Triglycerides From Baseline to Day 180
Description: LS mean percent change from baseline to Day 180 in Triglycerides in obicetrapib group compared to the placebo group
Time Frame: 180 Days
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 12.43 (4.178) | 4.49 (2.885)

20. Secondary Outcome: Precent Change in Triglycerides From Baseline to Day 365
Description: LS mean percent change from baseline to Day 365 in Triglycerides in obicetrapib group compared to the placebo group
Time Frame: 365 days
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10 mg
Number analyzed (Participants) | 118 | 234
percent change from baseline | 7.39 (5.642) | 2.27 (3.219)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 54
Description: Safety Population included all participants who received at least 1 dose of any study drug.
Arm/Group | Placebo | Obicetrapib 10 mg
All-Cause Mortality (participants affected / at risk) | 2/118 | 3/234
Serious Adverse Events (participants affected / at risk) | 8/118 | 13/234
Other Adverse Events (participants affected / at risk) | 52/118 | 95/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=118) | Obicetrapib 10 mg (N=234)
Death (General disorders) | 1 (1) | 0 (0) — Death from natural causes
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Sudden cardiac death (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=118) | Obicetrapib 10 mg (N=234)
Influenza (Infections and infestations) | 7 (7) | 21 (22)
COVID-19 (Infections and infestations) | 8 (8) | 15 (16)
Nasopharyngitis (Infections and infestations) | 5 (5) | 15 (17)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 12 (15)
Urinary tract infection (Infections and infestations) | 5 (5) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (8)
Diarrhea (Gastrointestinal disorders) | 8 (9) | 9 (10)
Blood creatine phosphokinase increased (Investigations) | 5 (6) | 3 (4)
Hypertension (Vascular disorders) | 8 (10) | 14 (14)
Fatigue (General disorders) | 7 (7) | 2 (2)
Headache (Nervous system disorders) | 6 (8) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or 12 months after completion of the study, whichever occurs first, Institution may publish the results of its study data. Institution and PI shall provide sponsor with an advance copy of any proposed communications at least 60 days prior and Sponsor shall have 60 days to review. Sponsor may request (a) the deletion of any Confidential Information, (b) reasonable changes, or (c) a delay for an additional period, not to exceed 90 days.

DOCUMENTS (2):
  • Study Protocol (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT05425745/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT05425745/SAP_001.pdf